CLINICAL TRIAL: NCT05831657
Title: Prevent It 2.0/Prevention to Reduce Incidence of Sexual Abuse by Reaching Individuals Concerned About Their Risk to Young People - An Internet Mediated Cognitive Behavioral Therapy to Reduce the Risk of Committing Child Sexual Abuse
Brief Title: Prevent It 2.0/PRIORITY - An iCBT to Reduce the Risk of Committing Child Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Royal Ottawa Mental Health Centre (Other); Johns Hopkins Bloomberg School of Public Health (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Universidade do Porto (Other)
Responsible Party: Principal Investigator, Christoffer Rahm, MD, PhD, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prevent It 2.0/PRIORITY
Record Dates: First submitted 2023-01-31; First posted 2023-04-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-10

CONDITIONS: Pedophilia
Keywords: Child sexual abuse; Pedophilic disorder; Preventive psychiatry; Internet based intervention; Cognitive behavioral therapy; Waitlist
MeSH Terms: conditions — Pedophilia | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: An academically initiated randomized controlled clinical trial where Prevent It 2.0 is compared with waitlist control across three language sites (i.e., Swedish, Portuguese, and German)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Prevent It 2.0 Swedish (Experimental): A free, anonymous, internet-delivered, clinician-guided, cognitive behavioral therapy (CBT) intervention delivered in Swedish.
  Interventions: Other: Prevent It 2.0
- Waitlist Swedish (Active Comparator): Waitlist Swedish Participants in the waitlist control will wait thirteen weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing problematic sexual behavior in Swedish.
  Interventions: Other: Waitlist
- Prevent It 2.0 German (Experimental): A free, anonymous, internet-delivered, clinician-guided, cognitive behavioral therapy (CBT) intervention delivered in German
  Interventions: Other: Prevent It 2.0
- Waitlist German (Active Comparator): Participants in the waitlist control will wait thirteen weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing problematic sexual behavior in German
  Interventions: Other: Waitlist
- Prevent It 2.0 Portuguese (Experimental): A free, anonymous, internet-delivered, clinician-guided, cognitive behavioral therapy (CBT) intervention delivered in Portuguese
  Interventions: Other: Prevent It 2.0
- Waitlist Portuguese (Active Comparator): Participants in the waitlist control will wait thirteen weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing problematic sexual behavior in Portuguese
  Interventions: Other: Waitlist

INTERVENTIONS:
Other: Prevent It 2.0 — A free, anonymous, internet-delivered, therapist assisted, cognitive behavioral therapy (CBT) intervention
  Arms: Prevent It 2.0 German; Prevent It 2.0 Portuguese; Prevent It 2.0 Swedish
Other: Waitlist — Participants in the waitlist control will wait thirteen weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing problematic sexual behavior.
  Arms: Waitlist German; Waitlist Portuguese; Waitlist Swedish

SUMMARY:
Child sexual exploitation and abuse is a large-scale global issue that has been drastically rising since the advent of the internet that has brought about communication technologies enabling new ways to sexually abuse children.

Prevent It is a free, anonymous, internet-delivered, and clinician-guided, cognitive behavioral therapy (CBT) intervention for adults who are concerned about their urges to engage in child sexual exploitation or abuse behaviors. It was developed based on many years of clinical experience from working with this patient group, as well as results from several previous research projects in the area of child sexual abuse.

Using a randomized controlled trial with waitlist control - a scientifically rigorous design - we will evaluate the effectiveness of the Swedish, German, and Portuguese versions of Prevent It 2.0 - an updated version of the initial Prevent It program. This evaluation is being funded by the European Commission and will consist of an international, multicentre, and academically initiated randomized controlled clinical trial for which those actively enrolled in Prevent It 2.0 will be compared to a waitlist control for each language version (Swedish, German, and Portuguese). Data will be collected across the three sites (Sweden, Germany, and Portugal), in their corresponding languages (Swedish, German, and Portuguese), over 18 months.

All data will be collected through the Iterapi platform that will be housed in a server by members of the Swedish subgroup located at Linköping University (LiU), Sweden. PRIORITY will provide intervention to 420 participants who will be recruited via multiple channels (darknet, Clearnet, police referral). Participation in the program will take place on both Darknet and Clearnet. All contact with participants, the treatment evaluations, and termination of the contact, is conducted via the online treatment platform Iterapi. The Iterapi platform is designed specifically for clinical trials of internet-mediated CBT.

DETAILED DESCRIPTION:
Child sexual exploitation and abuse is a large-scale global issue that has been drastically rising since the advent of the internet that has brought about communication technologies enabling new ways to sexually abuse children. In addition, existing programs for individuals concerned about their sexual urges and behavior toward children are generally sparse across the European Union (EU) and most have not been evaluated using rigorous scientific designs. Furthermore, those seeking to participate in prevention programs are often met with many internal and external barriers.

Therefore, to reduce the barriers often faced by those seeking help for their sexual urges to engage in child sexual exploitation or abuse, Prevent It was developed. Prevent It is a free, anonymous, internet-delivered, and clinician-guided, cognitive behavioral therapy (CBT) intervention for adults who are concerned about their urges to engage in child sexual exploitation or abuse behaviors. It was developed based on many years of clinical experience from working with this patient group, as well as results from several previous research projects in the area of child sexual abuse. Pilot results from a randomized clinical trial that assigned 160 child sexual abuse material (CSAM) users recruited from darknet forums to the intervention or placebo condition found that Prevent It significantly reduced CSAM use, that the program was safe from a negative side effects perspective, and well appreciated by the participants. However, the evaluation also revealed that participant attrition was high, particularly in the intervention condition, with almost half of the participants dropping out after the first two modules.

Prevent It was updated to Prevent It 2.0 based on feedback from participants and clinicians in the pilot study. It now contains 9 modules - with the first module focused on motivational engagement - that are completed over 9 weeks, with a 4 week follow up. The content of the therapy provided is classic CBT. Prevent It 2.0 will be provided in English, Swedish, German, and Portuguese. The Swedish, German, and Portuguese language versions are being evaluated within the framework of this project.

Using a randomized controlled trial with waitlist control - a scientifically rigorous design - we will evaluate the effectiveness of the Swedish, German, and Portuguese versions of Prevent It 2.0. This is part of a larger project (Prevention to Reduce Incidence of Sexual Abuse by Reaching Individuals Concerned About Their Risk to Young People; PRIORITY) funded by the European (EU) Commission aimed at translating and culturally adapting Prevent It 2.0 into German, Portuguese, and Swedish. Effectiveness of the program will be evaluated based on the impact of Prevent It 2.0 on participants sexual urges toward children.

Evaluating the efficacy of Prevent It 2.0 will consist of an international, multicentre, and academically initiated randomized controlled clinical trial for which those actively enrolled in Prevent It 2.0 will be compared to a waitlist control for each language version (Swedish, German, and Portuguese). Data will be collected across the three sites (Sweden, Germany, and Portugal), in their corresponding languages (Swedish, German, and Portuguese), over 18 months. All data will be collected through the Iterapi platform that will be housed in a server by members of the Swedish subgroup located at Linköping University (LiU), Sweden. PRIORITY will provide intervention to 420 participants who will be recruited via multiple channels (Darknet, Clearnet, police referral). Participation in the program will take place on both Darknet and Clearnet. All contact with participants, the treatment evaluations, and termination of the contact, is conducted via the online treatment platform Iterapi. The Iterapi platform is designed specifically for clinical trials of internet-mediated CBT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Concerned about sexual urges regarding children
* Informed consent to participate

Exclusion Criteria:

* Participants with a severe psychiatric illness (such as high acute suicide risk or severe substance abuse)
* Participants that are judged to have a limited understanding of the languages that the treatment is delivered in (German, Swedish, and Portuguese)
* Lack serious intention to participate (assessed by the researcher/clinician during the intake interview, which lasts approximately one hour)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Is Prevent It 2.0 effective in changing participants' urges to act on sexual behaviors involving children, as measured by the SSAS (Sexual Symptom Assessment Scale) across each language version? | At time of registration of the intervention, immediately before the intervention/pre-intervention, during the intervention up to 8 weeks, immediately after the intervention, and four weeks after the intervention
  SSAS; scores for each item range from 0 to 4; total scores range from 0 to 48; higher scores indicate a worse outcome [i.e., more sexual urges involving children]

SECONDARY OUTCOMES:
Is Prevent It 2.0 effective in changing participants' sexual behaviors involving children, as measured by the Sexual Child Molestation Risk Assessment (the SChiMRA+) Part B across each language version? | Immediately before the intervention/pre-intervention, during the intervention up to 8 weeks, immediately after the intervention, and four weeks after the intervention.]
  There's no scoring system at the moment. It's all item-by-item. But for all items, higher values indicate a worse outcome [e.g., more hours watching CSAM, etc.]
Is Prevent It 2.0 effective in changing participants' likelihood of engaging in sexual behaviors involving children, as measured by the Sexual Child Molestation Risk Assessment (the SChiMRA +) Part A across each language version? | Immediately before the intervention/pre-intervention, during the intervention up to 8 weeks, immediately after the intervention, and four weeks after the intervention.
  There's no scoring system at the moment. It's all item-by-item. But for all items, higher values indicate a worse outcome [e.g., more motivation to interact with children, etc.]

OTHER OUTCOMES:
Is Prevent It 2.0 effective in changing participants' acute dynamic risk of engaging in sexual behaviors involving children as measured by the Acute-2007-SR, across each language version? | During the intervention up to 8 weeks, and immediately after the intervention
  Acute-2007-Self-Report (i.e., self-report dynamic risk instrument based on the file coded Acute-2007; each item is scored as 0 = [no], 1 = [sometimes], and 3 = [often/frequently], with the exception of one item that is scored 0 = [no] and 1 = [yes]; total scores can range from 0 to 41; higher scores indicate a worse outcome [i.e., greater risk of engaging in sexual behaviors involving children]
Is Prevent It 2.0 effective in changing participants' sexual preoccupation, as measured by the Sexual Behavior Involving Minors Scale (SBIMS) - Part A across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  Each item is scored on a Likert scale from 1 = [never] to 5 = [daily]; total scores range from 4 to 20; higher scores indicate a worse outcome [i.e., more sexual preoccupation]
Is Prevent It 2.0 effective in changing participants' sexual self-control, as measured by the Hypersexual Behavior Inventory (HBI-19) - control and consequences items across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  Each item is scored on a Likert scale from 1 = [never] to 5 = [very often]; total scores each item is scored on a Likert scale from 1 = [never] to 5 = [very often]; total scores range from 12 to 60; higher scores indicate a worse outcome [i.e., less sexual self-control]
Is Prevent It 2.0 effective in changing participants' sexualized coping, as measured by the Hypersexual Behavior Inventory (HBI-19) - coping items across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  Each item is scored on a Likert scale from 1 = [never] to 5 = [very often]; total scores range from 7 to 35; higher scores indicate a worse outcome [i.e., more sexualized coping/using sex to cope]
Is Prevent It 2.0 effective in changing participants' emotional identification with children, as measured by the Child-like Sense of Self subscale of the Cognitive and Emotional Congruence with Children (C-ECWC) scale across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  Each item is scored on a Likert scale from 1 = [strongly disagree] to 4 = [strongly agree]; total scores range from 5 to 20; higher scores indicate a worse outcome [i.e., more emotional congruence with children]),
Is Prevent It 2.0 effective in changing participants' offense-supportive cognitions, as measured by the Sex With Children (SWCH) scale, across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  Each item is scored on a Likert scale from 0 = [strongly disagree] to 4 = [strongly agree]; total scores range from 0 to 32; higher scores indicate a worse outcome [i.e., more cognitions supportive of child sexual exploitation and abuse]
Is Prevent It 2.0 effective in changing participants' alcohol use, as measured by the Quantity-Frequency measure, across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  i.e., "About how often did you drink any alcohol in the past week/month?", item is scored from 0 = [did not drink any] to 4 = [7 days a week]; "Think of all of the times you had alcohol in the past week/month. When you drank alcohol, how much did you usually have at one time, on average during this week/month?", item is open ended response of number of glasses; higher scores indicate greater alcohol consumption
Is Prevent It 2.0 effective in changing participants' negative affect, as measured by the Patient Health Questionnaire, across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  PHQ-9; each item is scored on a Likert scale from 0 = [not at all] to 3 = [nearly every day]; total scores can range from 0 to 27; higher scores indicate a worse outcome [i.e., more negative affect]
Is Prevent It 2.0 effective in changing participants' motivation for change, as measured by the Readiness to Change Questionnaire, across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  Each item is scored on a Likert scale from -2 = [strongly disagree] to +2 = [strongly agree]; total scores for precontemplation, contemplation and action stages range from -4 to +4; higher scores indicate greater likelihood that the participant is in that stage of change
Is Prevent It 2.0 effective in changing how participants spend their leisure and recreation time, measured by having participants self-report to how they usually spend their leisure/recreation time, across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  i.e., "How do you usually spend most of your free time?" and "Who do you usually spend most of your free time with?"; respondent selects all category options that apply [e.g., categories include things like "doing sports, lazing around, watching television, etc."
Is Prevent It 2.0 effective in changing participants' social connection/loneliness, as measured by the Perceived Social Support Questionnaire, across each language version? | Immediately before the intervention/pre-intervention, immediately after the intervention, and four weeks after the intervention
  F-SozU K6; each item is scored on a Likert scale from 1 = [Note true at all/Does not apply] to 5 = [Very true/Exactly applicable]; total scores range from 6 to 30; higher scores indicate a better outcome [i.e., more perceived social support]
Is Prevent It 2.0 safe from a negative side effects perspective, as measured by the Negative Effects Questionnaire, across language version? | Immediately after the intervention
  NEQ-20; taps the occurrence [binary, yes or no] and severity [on a 5-point Likert scale 0-4, ranging from "not at all" to "extremely"] of 20 statements regarding negative effects of psychological treatment and ends with one free-text question. For each statement answered with yes , the respondent also reports whether they believe the negative effect is caused by "the treatment I received" or "other circumstances". Maximum score = 80, Minimum score = 0
Comparisons on participants' paraphilic interests, as measured by the Self-rating Sexual Interests (LASSIE) scale - version 2.1, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  Each item is scored on a Likert scale from 0 = [I disagree completely] to 3 = [I completely agree]; total scores range from 0 to 225; higher scores indicate more paraphilic interests
Comparisons on participants' criminal history, measured by self-reported prior charges related to violent, sexual, or non-violent criminal offences, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  i.e., "Have you ever been charged for a non-violent criminal offense, excluding minor traffic violations", "Have you ever been charged for a non-sexual violent offense", "Have you ever been charged for a non-contact sexual offense", and "Have you ever been charged for a contact sexual offense"; items are scored as dichotomous ratings of 1 = [yes] and 0 = [no]; higher scores indicate a worse outcome [i.e., more prior criminal charges]
Comparisons on participants' history of relationship instability, measured by self-reported items assessing historical relationship instability, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  i.e., "What is your current relationship status", for this item respondent selects all categorical responses that apply to their current relationship status [e.g., Married/ in a civil partnership and living together, Married/ in a civil partnership and not living together, In a steady relationship and living together, etc.]; "How many previous cohabitating romantic partner have you had?", for this item respondent selects 1, 2, 3, 4, 5, 6, or more; higher scores indicate more historical relationship instability
Comparisons on participants' history of employment/education instability, measured by participants' self-report to items assessing this, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  i.e., "Have you maintained stable employment or continued enrollment in educational studies over the last year leading up to your enrollment in this program", item is scored according to a dichotomous rating of 0 = [yes] and 1 = [no]; "Have you ever been unemployed or dropped out of school for a period of a year or more?", item is scored according to a dichotomous rating of 0 = [no] and 1 = [yes]; higher scores indicate a worse outcome [i.e., more historical education/employment instability]
Comparisons on participants' history of alcohol abuse, as measured by the Alcohol Use Disorders Identification Test - Consumption items, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  AUDIT-C; each item is scored from 0 to 4; total scores range from 0 to 12; higher scores indicate a worse outcome [i.e., more alcohol use/abuse]
Comparisons on religiosity/spirituality, measured by having participants' self-report to items assessing religious/ spiritual practices, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  i.e., "How important is religion/spirituality in your life?", item is scored on a Likert scale from 0 = [Not at all important] to 3 = [Very important]; "How often do you engage in religious/spiritual practice?", item is scored on a Likert scale from 0 = [Never] to 3 = [Every day]; higher scores indicate greater religiosity/spirituality
Comparisons on participants' adverse childhood experiences, as measured by the Adverse Childhood Experiences (ACEs) Questionnaire, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  Ratings of "yes" for dichotomous variables and ratings of "once or twice" to "very often" for frequency items are scored as 1 [exposed to ACE), while ratings of "no" or "never" are rated as 0 [not exposed], a domain is rated as 1 = "exposed to ACE" if the respondent indicates exposure to at least one item in that domain; total scores range from 0 to 8; higher scores indicate a worse outcome [i.e., greater exposure to adverse childhood experiences]
Comparisons on autism, as measured by the Ritvo Autism and Asperger Diagnostic Scale - 14-item Screener, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  RAADS-14; all items are scored from 0 to 3, total scores range from 0 to 42; higher scores indicate more autism spectrum symptoms
Comparisons on participants' engagement in prior child sexual abuse behaviors, as measured by the Sexual Behavior Involving Minor Scale (SBIMS) - Part B, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  Each item is scored on a Likert scale from 1 = [never] to 5 = [daily]; total scores range from 5 to 25; higher scores indicate a worse outcome [i.e., more prior child sexual abuse behaviors]
Comparisons on participants' static risk in relation to sexual abuse, as measured by self-reported items created out of the Static-99R, between active arm and waitlist in Prevent It 2.0 and between language versions will be conducted | At time of registration of the intervention
  i.e., a well-validated instrument for assessing static risk of sexual abuse that is usually file coded; total scores can range from -3 to 12; higher scores indicate greater risk of engaging in sexual abuse

CONTACTS AND LOCATIONS:
Overall Officials: Peer Briken, MD, Principal Investigator — Co-investigator, Universitaetsklinikum Hamburg-Eppendorf; Joana Carvalho, PhD, Principal Investigator — Co-investigator, Universidade Do Porto; Michael Seto, PhD, Principal Investigator — Co-investigator, The Royal Ottawa Health Care Group; Elizabeth J Letourneau, PhD, Principal Investigator — Co-investigator, Moore Center for the Prevention of Child Sexual Abuse
Locations (3):
- Universitaetsklinikum Hamburg-Eppendorf, Hamburg, Germany, Germany
- Universidade Do Porto, Porto, Praça de Gomes Teixeira, Portugal
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in each respective article, after deidentification (text, tables, figures, and appendices). Fully deidentified participant data will be shared in a public repository without demographic information. Data with demographic information will be shared with an approved data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For data shared through a data access agreement, beginning 3 months and ending 5 years following each article publication. Data shared in a public repository will be available immediately following each article publication and will be available for at least 5 years.
Access Criteria: For data that contain demographic information, investigators who provide a methodologically sound proposal, and whose proposed use of the data has been approved by an independent review committee identified for this purpose. Any researcher may access the version of the data available in a public repository.
  * For what types of analyses? To achieve aims in the approved proposal and for meta-analysis
  * By what mechanism will data be made available? Proposals should be directed to Christoffer.rahm@ki.se. To gain access to the data with demographic information, data requesters will need to sign a data access agreement. Data will be made available digitally via a secure data transfer facility provided by Karolinska Institute. Fully deidentified data without demographics will be made available on the Open Science Framework (osf.io).

REFERENCES:
- [Background] Latth J, Landgren V, McMahan A, Sparre C, Eriksson J, Malki K, Soderquist E, Oberg KG, Rozental A, Andersson G, Kaldo V, Langstrom N, Rahm C. Effects of internet-delivered cognitive behavioral therapy on use of child sexual abuse material: A randomized placebo-controlled trial on the Darknet. Internet Interv. 2022 Nov 15;30:100590. doi: 10.1016/j.invent.2022.100590. eCollection 2022 Dec. PMID 36573073